## DEVELOPMENT, VALIDATION, AND EVALUATION OF THE EFFECTIVENESS OF SIMULATION IN BASIC LIFE SUPPORT TRAINING (SBLST), ON NEWLY EMPLOYED NURSES IN GOVERNMENTAL JORDANIAN HOSPITALS

## **Consent Form**

Last update 0n 20-4-2023 Malaysian Human subjects protection review board date: 20-4-2023

\*

## Subject Information and Consent Form (Signature Page)

Research title: DEVELOPMENT, VALIDATION, AND EVALUATION OF THE EFFECTIVENESS OF SIMULATION IN BASIC LIFE SUPPORT TRAINING (SBLST), ON NEWLY EMPLOYED NURSES IN GOVERNMENTAL JORDANIAN HOSPITALS

Researcher's Name: Yousef Abu-Wardeh, Dr. Zakira Binti Mamat, Dr. Intan Idiana Binti Hassan

You or your legal representative must sign this page to participate in this study; by signing this page, I am confirming the following:

I have read all of the information in this Patient Information and Consent Form, including any information regarding the risk in this study, and I have had time to think about it.

All of my questions have been answered to my satisfaction. I voluntarily agree to be part of this research study, to follow the study procedures, and to provide necessary information to the doctor, nurses, or other staff members, as requested.

I may choose to stop participating in this study at any time.

I have received a copy of this Participant Information and Consent Form to keep.

| Participant Name | |
|-------------------------------------------------------|-----------------|
| Participant I.C No | |
| Signature of Participant or Legal Representative | Date (dd/MM/yy) |
| Name of Individual Conducting Consent Discussion | |
| Signature of Individual Conducting Consent Discussion | Date (dd/MM/yy) |
| Name & Signature of Witness (dd/MM/yy) | Date |

Note: i) All participants involved in this study will not be covered by insurance.

\*

## Participant's Material Publication Consent Form Signature Page

Research title: DEVELOPMENT, VALIDATION, AND EVALUATION OF THE EFFECTIVENESS OF SIMULATION IN BASIC LIFE SUPPORT TRAINING (SBLST), ON NEWLY EMPLOYED NURSES IN GOVERNMENTAL JORDANIAN HOSPITALS Researcher's Name: Yousef Abu-Wardeh, Dr. Zakira Binti Mamat, Dr. Intan Idiana Binti Hassan

You or your legal representative must sign this page to participate in this study.

By signing this page, I am confirming the following:

I understood that my name would not appear on the materials published, and there have been efforts to make sure that the privacy of my name is kept confidential, although confidentiality is not completely guaranteed due to unexpected circumstances.

I have read the materials or general description of the material and reviewed all photographs and figures I am included that could be published.

I have been offered the opportunity to read the manuscript and see all materials I am included in, but I have waived my right to do so.

All the published materials will be shared among medical practitioners, scientists and journalists worldwide.

The materials will also be used in local and book publications and accessed by many local and international doctors worldwide.

I, at this moment, agree and allow the materials to be used in other publications required by other publishers with these conditions:

The materials will not be used for advertising purposes nor as packaging materials.

The materials will not be used out of contex - i.e., Sample pictures will not be used in an article that is unrelated subject to the picture.

| Participant Name | | |
|-------------------------|-------------------------|-----------------|
| Participant I.C No. | Participant's Signature | Date (dd/MM/yy) |
| Name and Signature of I | ndividual | Date (dd/MM/yy) |

\*